CLINICAL TRIAL: NCT07209033
Title: A Prospective, Randomized, Double-blinded, Multi-center, Non-inferiority Study Evaluating the Efficacy, Safety and Long-term (Radiological and Clinical) Outcomes During Comprehensive Care Continuum of Implanted Biocomposite for Bone Regeneration FlexiOss® Compared to the Current Standard of Care in Patients With Primary Acute Trauma Bone Defects.
Brief Title: FlexiOss® - Efficacy, Safety and Long-term (Radiological and Clinical) Outcomes During Comprehensive Care Continuum of Implanted Biocomposite for Bone Regeneration.
Acronym: FlexiOssOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Inventi S.A. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-MED-0003
Record Dates: First submitted 2025-08-14; First posted 2025-10-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Bone Defect
Keywords: Bone Defect; Bone Trauma; Bone Injury; Biocomposite; Bone Regeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The trial is double-blinded, keeping sponsor, all patients and the assessors blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone reconstruction with FlexiOss® biocomposite (Experimental)
  Interventions: Device: FlexiOss®
- Control group with allogenic human bone grafting (Active Comparator)
  Interventions: Procedure: Allogenic human bone grafting

INTERVENTIONS:
Device: FlexiOss® — Bone reconstruction with FlexiOss® biocomposite.
  Arms: Bone reconstruction with FlexiOss® biocomposite
Procedure: Allogenic human bone grafting — Implantation of allogenic human bone graft.
  Arms: Control group with allogenic human bone grafting

SUMMARY:
The aim of this clinical study is to evaluate the efficacy, safety and long-term (radiological and clinical) outcomes during comprehensive care continuum of implanted biocomposite for bone regeneration FlexiOss® compared to the current standard of care in patients with primary acute trauma bone defects.

The efficacy, safety and long-term (radiological and clinical) evaluation will be assessed during follow up visits at 2, 6 weeks, 3, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years.
2. Subject signed informed consent form and is willing to participate in the follow-up visits.
3. Subject with an existing acute primary bone defect in one of the following groups:

   1. Long bones of the lower extremity (including articular tibia plateau acute fracture).
   2. Bones of the foot (including articular calcaneus acute fracture).
4. Subject scheduled for orthopedic procedure with bone substitute material.

Exclusion Criteria:

1. Subject with alcohol dependence syndrome or any history of substance abuse within the past year.
2. Pregnancy or breastfeeding.
3. Subject participates in another clinical trial.
4. Unstable mental condition or psychiatric concomitant disease.
5. Diagnosed severe degenerative, metabolic bone disease or any condition that in opinion of the Investigator could adversely affect bone healing and regeneration.
6. Subject with known allergies or hypersensitivity to any components of the FlexiOss® biocomposite material
7. Subject with active cancer disease and/or during related oncological treatment.
8. Contraindications for computed tomography angiography according to the site Standard of Care include, but are not limited to, allergic reactions to contrast agents and impaired renal function.
9. Subject with severe comorbidities that could interfere with the study outcomes or pose a risk during surgery and rehabilitation.
10. Any other condition precluding implantation of FlexiOss®.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint | At 24-month follow-up
  Presence of bone union with maintained anatomic alignment and stable fixation, including support of the joint surface with a material capable of bone remodelling, as assessed by X-ray or CT at 24 months.
Number and Frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 24 months
  To measure the number and frequency of adverse event(s) (AEs) including serious adverse event(s) (SAEs) throughout the 24 months study duration.
Improvement of load-bearing capacity with simultaneously reduction of lower extremity dysfunction in the period before and after rehabilitation based on a PROMs (LEFS scale) over 24 months | At 2-week, 6-week, 3-month, 6-month, 12-month & 24-month follow-up
  To assess the improvement of load-bearing capacity and reduction of lower extremity dysfunction in the period before and after rehabilitation. The assessment is based on a Patient-Reported Outcome Measure (PROM), specifically the Lower Extremity Functional Scale (LEFS). The LEFS score ranges from 0 to 80, where a higher score indicates a better functional outcome.
Non-deterioration in Quality of Life (QoL) after completing rehabilitation based on SF-36 questionnaire score. | Up to 24 months
  To assess the non-deterioration in Quality of Life (QoL) using the MOS 36-item Short-Form Health Survey (SF-36). The scores for each domain of the SF-36 are transformed to a scale from 0 to 100, where a higher score indicates a better health outcome.

SECONDARY OUTCOMES:
Lack of reinterventions in the treated area within 24 months. | Up to 24 months
Full load on the treated limb during physical examination (lower limb bones) at 2 and 6 weeks; 3, 6, 12 and 24 months. | At 2 and 6 weeks; 3, 6, 12 and 24 months
  The ability to bear full load on the treated limb is assessed by an experienced orthopedist during scheduled study follow-up visits. The assessment is based on a physical examination where the physician's documented clinical judgment is determined by observing the patient's gait and ability to stand on the treated limb without assistance.
Full mobility of the treated limb during physical examination expressed as active or passive range of motions specific to the studied region at 2 and 6 weeks; 3, 6, 12 and 24 months. | At 2 and 6 weeks; 3, 6, 12 and 24 months
Lack of bone lysis in X-ray after 12 and 24 months (preserving joint surface alignment). | After 12 and 24 months
Assessment of changes in levels of calcium in blood after biocomposite implantation during follow-up at screening, 6 weeks, 6, 12, 24 months. | At screening, 6 weeks, 6, 12, 24 months
  The unit of measure will be reported in mg/dL.
Assessment of changes in levels of phosphates in blood after biocomposite implantation during follow-up at screening, 6 weeks, 6, 12, 24 months. | At screening, 6 weeks, 6, 12, 24 months
  The unit of measure will be reported in IU/L.
Proper bone union observed in imaging examination (X-ray) after 6 and 12 months. | After 6 and 12 months
Assessment of PROM - LEFS obtained individual results at discharge; 2 and 6 weeks; 3, 6, 12 and 24 months. | At baseline; 2 and 6 weeks; 3, 6, 12 and 24 months
  The specific PROM assessed here is the Lower Extremity Functional Scale (LEFS). The score ranges from 0 to 80, where a higher score indicates better functional ability. The baseline assessment for this measure is performed at the time of discharge from the hospital.
Assessment of PROM - SF-36 obtained individual results at discharge; 2 and 6 weeks; 3, 6, 12 and 24 months. | At baseline; 2 and 6 weeks; 3, 6, 12 and 24 months
  The specific PROM assessed here is the SF-36 Health Survey. The scores for each domain are transformed to a scale from 0 to 100, where a higher score indicates a better health outcome. The baseline assessment for this measure is performed at the time of discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Kamiński, Professor, Principal Investigator — Samodzielny Publiczny Szpital Kliniczny im. prof. Adama Grucy CMKP; Amadeusz Skiba, PhD, Principal Investigator — 5 Wojskowy Szpital Kliniczny z Polikliniką SP ZOZ
Locations (2):
- Poland (2):
  - Klinika Chirurgii Urazowej i Ortopedii 5 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Krakow
  - Klinika Chirurgii Urazowej Narządu Ruchu i Ortopedii CMKP Samodzielny Publiczny Szpital Kliniczny im. prof. Adama Grucy Centrum Medycznego Kształcenia Podyplomowego, Otwock

IPD SHARING:
Plan to Share IPD: No